CLINICAL TRIAL: NCT01561027
Title: A Randomized, Double Blind, Cross-over Study to Evaluate the Safety and Efficacy of CNV1014802 in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Crossover Study of CNV1014802 in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CNV1014802/201
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Lumbosacral Radiculopathy
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNV1014802 (Experimental): CNV1014802 350mg on prescription (BID) for 21 days
  Interventions: Drug: CNV1014802
- Placebo (Placebo Comparator): Placebo 350mg BID for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNV1014802 — Administered as specified in treatment arm.
  Arms: CNV1014802
Drug: Placebo — Administered as specified in treatment arm
  Arms: Placebo

SUMMARY:
The study is a randomized, double blind, cross-over study to evaluate the safety and efficacy of CNV1014802 in subjects with neuropathic pain from lumbosacral radiculopathy.

DETAILED DESCRIPTION:
The study consists of two treatment periods of 22 days with randomized CNV1014802 350mg or placebo administered twice daily. In addition, single blind placebo will be administered during a two week run-in, a two week wash-out period between the two treatment periods, and a one week run-out phase.

This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged between 18 and 65 years, with a diagnosis of neuropathic pain due to lumbosacral radiculopathy (LSR).
* Female subjects must be of non-child bearing potential or agree to use an approved form of contraception
* Body weight < 50 kg for men and < 45 kg for women.
* Capable of giving written informed consent.
* Approved concomitant medications must have been stable for at least 4 weeks prior to day 1.
* Average baseline daily pain score for neuropathic pain due to LSR on the 11-point numerical rating scale of 4 or greater.

Key Exclusion Criteria:

* Subjects who are unable to reliably delineate or assess their own pain by anatomical location/distribution.
* Subjects with lumbar canal stenosis in which the pain in the lower limbs occur solely on walking and not at rest.
* Subjects with causes for their neuropathic pain other than LSR.
* Subjects who have received nerve blocks and/or steroid injections for neuropathic pain within 4 weeks prior to day 1.
* Subjects who are indicated for surgical treatment of lumbosacral radiculopathy.
* A positive pre-study drug screen.
* A positive history of HIV.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of any liver disease within the last 6 months, with the exception of known Gilbert's disease.
* History of excessive regular alcohol consumption within 6 months of the study.
* Subjects with a history or risk of seizures or a history of epilepsy, head injury or related neurological disorders
* Subjects with a history of uncontrolled or poorly controlled hypertension, with systolic BP frequently exceeding 160mmHg and/or diastolic BP frequently exceeding 100mmHg, or subjects who have BP greater than or equal to 160mmHg systolic and/or greater than or equal to 100mmHg diastolic at screening after repeated measurements
* History or presence of significant cardiovascular, gastro-intestinal, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Subjects with conditions known to affect cardiac conduction or a personal or familial history of Brugada syndrome
* Pregnant females or lactating females.
* History or presence of any clinically significant abnormality in vital signs / ECG / laboratory tests or have any medical or psychiatric condition, which, in the opinion of the Investigator may interfere with the study procedures or compromise subject safety.
* History of suicidal ideation and/or suicide attempts or clinical evidence of recent major depression.
* Subjects who are unable to maintain their same medications for the treatment of neuropathic pain at a stable dose during the study.
* Unable to refrain from excessive use of sedatives.
* Unable to comply with the prohibited concomitant medication restrictions as detailed in the protocol. This includes but is not limited to sodium channel blockers or drugs that adversely interact with a monoamine oxidase-B inhibitor: MAOI's, antidepressants, opioids and sympathomimetic agents.
* Unable to stop and remain abstained from non-pharmacological treatments for their neuropathic pain during the study.
* History of hypersensitivity to CNV1014802.
* The subject has participated in a clinical trial and has received an investigational product within 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the start of this study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subject is mentally or legally incapacitated.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Neuropathic Pain Score from Baseline | Three weeks
  Change in average daily neuropathic pain score from baseline (average days 10-14) to week 3 based on the 11 point Pain Intensity Numerical Rating Scale (PI-NRS) (0=no pain, 10=maximum pain imaginable).
  Subjects should specifically rate the pain intensity for the neuropathic pain associated with lumbosacral radiculopathy and not pain from other concomitant causes

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | 3 weeks
  Change in average daily pain score from baseline (average days 10-14) to week 1 and week 2 of treatment and 1 week following the end of randomized treatment.
Responder Rate | 3 weeks
  Proportion of patients who have >= 30% and >=50% reduction in average daily pain score relative to baseline during weeks 1, 2 and 3 of treatment and 1 week following the end of randomized treatment.
Galer Neuropathic Pain Scale | 3 weeks
  Change in Galer Neuropathic Pain Scale from baseline to week 3 of treatment.
Oswestry Disability Index | 3 weeks
  Change in average disability score from baseline to week 1, week 2 and week 3 of treatment based on Oswestry Disability Index
PGIC | 3 weeks
  Proportion of patients who have "improved", "much improved" or "very much improved" relative to baseline on the Patient Global Impression of Change (PGIC) on week 3 of treatment.
CGIC | 3 weeks
  Proportion of patients who have "improved", "much improved" or "very much improved" relative to baseline on the Clinical Global Impression of Change (CGIC) on week 3 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- Czechia (3):
  - Research Site, Brno
  - Research Site, Litoměřice
  - Research Site, Prachatice
- Denmark (2):
  - Research Site, Glostrup Municipality
  - Research Site, Odense
- France (4):
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Saint-Etienne
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm